CLINICAL TRIAL: NCT04024423
Title: Healthcare-associated Links in Transmission of Nontuberculous Mycobacteria Among Patients With Cystic Fibrosis
Brief Title: Healthcare-associated Links in Transmission of Nontuberculous Mycobacteria in Cystic Fibrosis
Acronym: HALTNTM
Status: Completed | Type: Observational
Sponsor: National Jewish Health (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Principal Investigator, Jane Gross, Assistant Professor, National Jewish Health
Other Study IDs: HS-3175
Record Dates: First submitted 2019-07-15; First posted 2019-07-18 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-12

CONDITIONS: Cystic Fibrosis; Nontuberculous Mycobacterium Infection
MeSH Terms: conditions — Cystic Fibrosis; Mycobacterium Infections, Nontuberculous

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Sputum samples of nontuberculous mycobacteria
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Related M. abscess isolates: Characterize the source(s) of direct or indirect patient-to-patient transmission of NTM within an individual CF healthcare setting among participants with highly related isolates.
  Interventions: Other: Epidemiologic investigation
- Unrelated M. abscessus isolates: Characterize the source(s) of direct or indirect patient-to-patient transmission of NTM within an individual CF healthcare setting among participants with unrelated isolates.
  Interventions: Other: Epidemiologic investigation
- Related M. avium isolates: Characterize the source(s) of direct or indirect patient-to-patient transmission of NTM within an individual CF healthcare setting among participants with highly related isolates.
  Interventions: Other: Epidemiologic investigation
- Unrelated M. avium isolates: Characterize the source(s) of direct or indirect patient-to-patient transmission of NTM within an individual CF healthcare setting among participants with unrelated isolates.
  Interventions: Other: Epidemiologic investigation
- Related M. intracellulare isolates: Characterize the source(s) of direct or indirect patient-to-patient transmission of NTM within an individual CF healthcare setting among participants with highly related isolates.
  Interventions: Other: Epidemiologic investigation
- Unrelated M. intracellulare isolates: Characterize the source(s) of direct or indirect patient-to-patient transmission of NTM within an individual CF healthcare setting among participants with unrelated isolates.
  Interventions: Other: Epidemiologic investigation

INTERVENTIONS:
Other: Epidemiologic investigation — Identification of overlaps in source(s) of care between participants with NTM isolates in a Cystic Fibrosis Care Center.

SUMMARY:
Sources of NTM infection and modes of transmission among CF patients are poorly understood. Healthcare-associated transmission of NTM among CF patients has been suspected and is of growing concern for CF Centers. There is a need for a systematic evidence-based approach to investigating potential episodes of healthcare-associated transmission. Clusters of highly similar strains of NTM in CF patients cared for at the same CF Center may arise from healthcare sources including patient-to-patient transmission and/or acquisition from water sources within a healthcare setting. The primary objective of the study is to facilitate a standardized process by which CF Centers may perform data abstraction on patients identified with highly similar NTM isolates and determine if clustered NTM strains are related to strains isolated from healthcare setting water biofilm sources. HALT NTM is available to the entire CF Foundation Care Network, under a collaborative agreement, to initiate a standardized, independent, confidential, internal NTM outbreak investigation. Patients that are identified by whole genome sequencing as having highly similar NTM strains and receiving care in the same CF Care Center are eligible. The study's primary endpoint is to identify potential modes and sources of healthcare-associated acquisition of CF NTM, thereby revealing risk factors for NTM acquisition.

ELIGIBILITY:
Inclusion Criteria:

* Participants with cystic fibrosis and respiratory NTM growth on one or more occasions

Exclusion Criteria:

* Participants without cystic fibrosis
* Participants without pulmonary NTM growth

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with cystic fibrosis and growth of respiratory NTM on one or more occasion that have undergone whole genome sequencing of the NTM core genome at National Jewish Health.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Number of cystic fibrosis participants with NTM isolates in related clusters and receiving care in the same Cystic Fibrosis Care Center as assessed by whole genome sequencing | Three years
  Retrospective epidemiologic study
Number of cystic fibrosis participants with NTM isolates matching environmental isolates from the participant's Cystic Fibrosis Care Center as assessed by whole genome sequencing | Three years
  Retrospective epidemiologic study

CONTACTS AND LOCATIONS:
Overall Officials: Jane E Gross, MD PhD, Study Director — National Jewish Health
Locations (1):
- National Jewish Health, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available to other researchers.

REFERENCES:
- [Derived] Gross JE, Caceres S, Poch K, Hasan NA, Davidson RM, Epperson LE, Lipner E, Vang C, Honda JR, Strand M, Strong M, Saiman L, Prevots DR, Olivier KN, Nick JA. Healthcare-associated links in transmission of nontuberculous mycobacteria among people with cystic fibrosis (HALT NTM) study: Rationale and study design. PLoS One. 2021 Dec 20;16(12):e0261628. doi: 10.1371/journal.pone.0261628. eCollection 2021. PMID 34929010

DOCUMENTS (1):
  • Study Protocol (2020-05-08): https://cdn.clinicaltrials.gov/large-docs/23/NCT04024423/Prot_000.pdf